CLINICAL TRIAL: NCT04183400
Title: Safety Awareness For Empowerment (SAFE): An RCT With Young People Experiencing Homelessness
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kimberly Bender, Professor, University of Denver
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UDenverSAFE; 1R15DA039355-01 (NIH)
Record Dates: First submitted 2019-11-15; First posted 2019-12-03 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Substance Use; Victimization
Keywords: substance use; victimization; homeless youth; youth experiencing homelessness
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Awareness For Empowerment (SAFE) (Experimental): Brief mindfulness-based cognitive-behavioral skill-building intervention
  Interventions: Behavioral: Safety Awareness For Empowerment (SAFE)
- Usual case management only (No Intervention): Control condition receives only services as usual

INTERVENTIONS:
Behavioral: Safety Awareness For Empowerment (SAFE) — SAFE is a mindfulness-based cognitive-behavioral intervention that aims to build risk-related attention skills.
  Arms: Safety Awareness For Empowerment (SAFE)

SUMMARY:
The SAFE study examines the effects of brief mindfulness-based cognitive-behavioral intervention aimed at improving risk-related attention skills (risk detection, problem solving, assertiveness, and help seeking) in order to reduce substance use and victimization among young people (ages 18-21) experiencing homelessness.

DETAILED DESCRIPTION:
Youth (ages 18-21) living at a local youth shelter will be recruited and randomly assigned to receive the SAFE intervention (plus usual case management) or to receive usual case management only. Those assigned to SAFE will receive 12 mindfulness-based, cognitive-behavioral modules through a 3-day intensive group intervention provided by an agency intern and a hired project staff member. The intervention uses mindfulness-based cognitive-behavioral approaches to augment youth attention to risk-related processes, including risk detection, problem solving, assertiveness, and help seeking skills. It is hypothesized the intervention will result in reduced substance use and victimization and that these effects will be explained, at least in part, by improved risk-related attention skills (risk detection, problem solving, assertiveness, and help seeking skills). Post baseline interview, participants will be randomly assigned and will participate in a posttest interview (1 week post baseline) and follow up interviews at 6-weeks, 3-months, and 6-months post baseline interview.

ELIGIBILITY:
Inclusion Criteria:

* Reside at the partnering community based youth shelter

Exclusion Criteria:

As measured by the KSADS (a semi-structured diagnostic interview administered by trained interviewers at baseline):

* presence of psychotic symptoms;
* presence of a life-threatening medical/chronic neurological illness that would prevent participation in a 4-day intervention and/or assessments;
* suicide attempt in last 6 months without current enrollment in therapy or related services to address;
* chronic self-injurious behavior/cutting without current enrollment in therapy or related services to address
* hospitalization or residential treatment for psychiatric reasons in last 6 months without current enrollment in therapy or related services to address.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Substance use | Follow up at 6-weeks post baseline interview
  The Substance use domain of the Addiction Severity Index, 5th edition will be used to assess the frequency, type and amount of substance use in the past 30 days. This domain will be adapted to add smoking tobacco to the list of substances.
Substance use | Follow up at 3-months post baseline interview
  The Substance use domain of the Addiction Severity Index, 5th edition will be used to assess the frequency, type and amount of substance use in the past 30 days. This domain will be adapted to add smoking tobacco to the list of substances.
Substance use | Follow up at 6-months post baseline interview
  The Substance use domain of the Addiction Severity Index, 5th edition will be used to assess the frequency, type and amount of substance use in the past 30 days. This domain will be adapted to add smoking tobacco to the list of substances.
Victimization | Follow up at 6-weeks post baseline interview
  The Juvenile Victimization Questionnaire (JVQ) will be used to asses exposure to a range of types of victimization.
Victimization | Follow up at 3-months post baseline interview
  The Juvenile Victimization Questionnaire (JVQ) will be used to asses exposure to a range of types of victimization.
Victimization | Follow up at 6-months post baseline interview
  The Juvenile Victimization Questionnaire (JVQ) will be used to asses exposure to a range of types of victimization.

SECONDARY OUTCOMES:
Substance use symptoms | Follow up at 6-weeks, 3-months, and 6-months post baseline interview, controlling for baseline
  The Mini International Neuropsychiatry Interview (MINI) will be used to assess a count of the number of substance use symptoms experienced.
Substance use disorder diagnostic criteria | Follow up at 6-weeks, 3-months, and 6-months post baseline interview, controlling for baseline
  The Mini International Neuropsychiatry Interview (MINI) will be used to assess a whether the participant meets DSM diagnostic criteria for a substance use disorder
Risk detection | Follow up at 1-week, 6-weeks, and 3-months post baseline interview, controlling for baseline
  Risk detection will be assessed a set of researcher-developed Risk Vignettes that describe characters in risk situations and ask participants to identify risk cues present; measure will be proportion of risk cues identified among those present in the vignettes administered
Help seeking intentions | Follow up at 1-week, 6-weeks, and 3-months post baseline interview, controlling for baseline
  Help seeking intentions will be assessed with a modified version of the General Help Seeking Questionnaire which assesses intentions to seek help from different sources for different problems. The original scale asks about seeking help for emotional problems and suicidal thoughts; our version was modified to ask about help seeking related to safety issues and substance use. Higher scores indicate greater help seeking thus a more positive outcome.
Help seeking behaviors | Follow up at 1-week, 6-weeks, and 3-months post baseline interview, controlling for baseline
  Help seeking behaviors will be assessed by items from the Help Seeking Behaviors scale which ask how often youth actually sought help fro different sources of help for substance and for safety.
Assertiveness | Follow up at 1-week, 6-weeks, and 3-months post baseline interview, controlling for baseline
  Assertiveness will be assessed using the Assertion Inventory which asks how often participants engage in assertive behaviors across three domains: substance use, general, and social situations

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Bender, PhD, Principal Investigator — University of Denver
Locations (1):
- Urban Peak Shelter and University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No